CLINICAL TRIAL: NCT03547050
Title: Rolandic Epilepsy Genomewide Association International Study
Acronym: REGAIN
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Cardiff University (Other); The Hospital for Sick Children (Other); Hospital JP Garrahan (Other Government); Aghia Sophia Children's Hospital of Athens (Other); Hospital Mutua de Terrassa (Other); Seattle Children's Hospital (Other); Hasbro Children's Hospital (Other); Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: 229844; TWF 164-3020 (Other Grant/Funding Number: The Waterloo Foundation)
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-03

CONDITIONS: Rolandic Epilepsy
Keywords: Epilepsy; Rolandic; Genetics; Genomewide Association Study; RE; Neurology; Pediatrics
MeSH Terms: conditions — Epilepsy, Rolandic; Epilepsy | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients diagnosed with RE: People who meet the eligibility requirements and have been diagnosed with rolandic epilepsy.
  Interventions: Other: Blood draw
- Controls: People without a lifetime history of seizures.
  Interventions: Other: Existing samples

INTERVENTIONS:
Other: Blood draw — Participation includes one visit for one blood draw per recruited patient. 10-20ml peripheral venous blood will be taken from the antecubital fossa. The DNA from the blood sample will then be extracted and resequenced for analysis.
  Groups: Patients diagnosed with RE
Other: Existing samples — Control DNA samples will be used that have been previously acquired in other studies.
  Groups: Controls

SUMMARY:
We have discovered a small change in the genetic code which increases the risk of the brainwave abnormality that is found in rolandic epilepsy. We now wish to confirm this using a second much larger sample of patients. We will investigate the other genetic changes that cause people with the brainwave abnormality to develop seizures, as well as problems with speech, coordination, attention and learning.

DETAILED DESCRIPTION:
Epilepsy is a common neurological disorder affecting 1% of the population. There are over 30 types of epilepsy, some common, some rare. Most epilepsies arise in childhood and have a genetic cause. Approximately 25% of child patients have "Rolandic Epilepsy" or RE, also known as Benign Epilepsy with Centrotemporal Spikes (BECTS). RE has a complex genetic basis, probably made up of combinations of susceptibility variants in different genes. Children with RE quite often have other symptoms that affect their speech, attention, reading ability or coordination. The goal of this study is to find the genetic basis for susceptibility to seizures and associated comorbidities for RE using genomewide association approaches.

We know that RE has a genetic basis and we recently discovered the genetic cause of the EEG pattern seen in RE. The goal of REGAIN is to now find the genetic basis for susceptibility to seizures and the associated symptoms above. Our hope is to be able to improve diagnosis and understand why each child with RE is different, and perhaps point us towards new treatments that are more effective and have fewer side effects.

We will compare the genetic code of 3,000 children with RE against a similar number of people not affected by epilepsy. With the proposed large sample of participants, we will be able to pinpoint the exact changes that might lead to seizures or attention problems for example. Learning the genetic basis for these problems will deepen our understanding of the mechanisms and lead to new treatments or cures.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Rolandic Epilepsy in accordance with the following international criteria:

   * Age of first afebrile seizure 3-12 years
   * Seizures comprising focal sensorimotor seizures affecting the vocal tract and face, with or without involvement of the arm
   * Predominant sleep-related seizures
   * EEG interictal centro-temporal spikes with normal background
2. Current age 6-25 years

Exclusion Criteria:

1. No history of focal seizure
2. Normal EEG or abnormal background features on EEG
3. Known structural causes (stroke, tuberous sclerosis, infection, post-infectious or metabolic)
4. Primary diagnosis of autism or global learning disability
5. Focal central neurological deficit on clinical exam,
6. Unable to provide informed consent
7. Unable to provide blood sample

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Target population is 3,000 participants with a diagnosis of Rolandic Epilepsy (1,000 UK).
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Allelic association p value corrected for genome wide testing | Day 1
  We will look to see if there are changes in the genetic code that cause brainwave abnormalities close to the genetic changes that we have already discovered.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (3):
  - Columbia University Medical Center, New York, New York
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Seattle Children's Hospital, Seattle, Washington
- Dr. Juan P. Garrahan Children's Hospital, Buenos Aires, Argentina
- Hospital for Sick Kids, Toronto, Ontario, Canada
- Aghia Sophia Children's Hospital of Athens, Athens, Greece
- Italy (2):
  - Sicilian Epilepsy Network, Catania
  - Commissione Genetica Lega Italiana contro l'Epilepssia, Roma
- Hospital Mutua de Terrassa, Barcelona, Spain
- United Kingdom (4):
  - Cardiff University School of Medicine, Cardiff
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Swansea University College of Medicine, Swansea

REFERENCES:
- See also: Childhood Epilepsy website — http://childhoodepilepsy.org